CLINICAL TRIAL: NCT06036537
Title: Investigation on Risk Factors of Rheumatoid Arthritis Related Interstitial Lung Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xiaocheng Cheng, M.D., First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 1stChongqingMU123
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis Associated Interstitial Lung Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- rheumatoid arthritis
  Interventions: Diagnostic Test: diagnosis of Interstitial lung disease

INTERVENTIONS:
Diagnostic Test: diagnosis of Interstitial lung disease — Serum marker detection，High resolution computed tomography scan

SUMMARY:
Rheumatoid arthritis (RA) is one of the most common autoimmune diseases, characterized by chronic inflammatory bone and cartilage destruction. Although treatment including anti-tumor necrosis factor (TNF) and interleukin-6 (IL-6) receptor antibodies has been successful, only 20% to 30% of patients have achieved complete remission. Interstitial lung disease (ILD) is a common complication of rheumatoid arthritis (RA). Approximately 5-10% of RA patients have clinically significant rheumatoid arthritis associated interstitial lung disease (RA-ILD), with a mortality rate of 2-10 times that of RA-non ILD patients. The median survival after diagnosis is between 3-8 years. Although there are multiple biomarkers for RA-ILD, such as anti citrullinated protein antibody (ACPA), MUC5B mutant gene, KL-6, etc., none of these biomarkers can reliably predict the disease and prognostic risk of RA-ILD. Therefore, improving the prediction of RA complicated with ILD and exploring risk factors for the progression and prognosis of RA-ILD can contribute to early diagnosis and treatment, and is of great significance in preventing RA lung injury and death.

This study aims to screen differential serum biomarkers between RA patients and RA-ILD patients through prospective cohort studies, to explore whether these differential serum biomarkers are a risk factor for RA patients complicated with ILD, and whether they affect the clinical prognosis of RA-ILD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of rheumatoid arthritis patients based on the 2010 ACR/EULAR RA classification criteria; 2. age ≥18 years; 3. Interstitial lung disease was diagnosed by lung high resolution computed tomography (HRCT)

Exclusion Criteria:

1. age <years; 2. Being treated with urate-lowering medications; 3. Other systemic/organ specific autoimmune diseases other than rheumatoid arthritis (such as SLE, ANCA associated vasculitis, pSS, SSc, myositis, etc.); 4.Tumor, pulmonary tuberculosis, glomerular filtration rate less than 30ml/min/1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: rheumatoid arthritis patients
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of interstitial lung disease | 2 years
  Whether rheumatoid arthritis patients have occurred interstitial lung disease and the time of occurrence of interstitial lung disease

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing General Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu Q, Cheng X, Lan Y, Lei H, Niu C, Luo Y. Serum uric acid predictive value and prognostic impact in rheumatoid arthritis' associated interstitial lung disease. Front Med (Lausanne). 2025 Aug 5;12:1623557. doi: 10.3389/fmed.2025.1623557. eCollection 2025. PMID 40837562